CLINICAL TRIAL: NCT05751382
Title: 3-year Evaluation of the Clinical Performances of a Self-adhesive Hybrid Resin Composite Compared to a Traditional Composite Resin Used for Direct Restorations of Non-carious Cervical Lesions (NCCLs): A Split-mouth Randomized Clinical Trial
Brief Title: Evaluation of Self-adhesive Hybrid Resin Composite Compared to a Traditional Composite Resin in Restorations of NCCLs
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to slow recruitment.
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14.1535
Record Dates: First submitted 2023-02-07; First posted 2023-03-02 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-11

CONDITIONS: Tooth Restoration

STUDY DESIGN:
Intervention Model Description: Split-mouth design, i.e. each subject have both treatment arms.
Who Masked: Outcomes Assessor
Masking Description: The aesthetic integration of the restoration will be evaluated by two experienced and blinded operators following the aesthetic criteria of the FDI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Restoration with Surefil one hybrid composite (Experimental): In a split-mouth design, subjects were randomly assigned to restoration with Surefil one hybrid composite in either the left or the right upper quadrant.
  Restoration performed with Surefil one hybrid composite applied according to manufacturer's instruction and cured for 20 seconds with a LED lamp (Smartlamp Pro).
  Interventions: Device: Surefil one
- Restoration with Venus Pearl composite (Active Comparator): In a split-mouth design, subjects were randomly assigned to restoration with Venus Pearl composite in either the left or the right upper quadrant.
  After the application of the adhesive system (iBond universal), the Venus Pearl composite will be layered on the cavity and cured for 20 seconds with a LED lamp Smartlamp Pro).
  Interventions: Device: Venus Pearl

INTERVENTIONS:
Device: Surefil one — Restorative material (Dentsply Sirona). Used for direct restoration of class V NCCL.
  Arms: Restoration with Surefil one hybrid composite
Device: Venus Pearl — Restorative material. Traditional paste composite employed in combination with iBond universal adhesive.
  Arms: Restoration with Venus Pearl composite

SUMMARY:
This is a split-mouth randomized clinical investigation conducted to evaluate clinical performances of a self-adhesive hybrid resin composite (investigational medical device Surefil) compared to a traditional composite resin, when used for direct restorations of non-carious lesions (NCCLs). The study consists of a 3-year long follow-up period.

DETAILED DESCRIPTION:
The aim of this study is to demonstrate non-inferiority in terms of clinical performance and patient discomfort after direct restorative treatment of class V NCCL with Surefil one restorative material (Dentsply Sirona) in combination with a traditional paste composite "Venus Pearl" employed in combination with iBond universal adhesive (Kulzer Dental) during an observational period of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients aging from 18 to 70
* 40-60% women, 40-60% men
* Patients who present at least 2 cervical lesions on canines and / or upper premolars on vital teeth
* Patients who are not allergic or sensitive to the ingredients contained in the products
* The test patient consents to the restorative treatment in line with the study´s criteria (informed consent)
* Sufficiently understanding of the language

Exclusion Criteria:

* Extremely low level of oral hygiene
* Teeth with previous restorations
* Not possible adequate isolation of the operating area
* Patients with serious systemic diseases
* Devitalized teeth or with pulpitis in progress
* Periodontal problems on the elements to be restored

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Breschi, Prof, Principal Investigator — Clinica Odontoiatrica (DIBINEM)
Locations (1):
- Clinica Odontoiatrica (DIBINEM), Bologna, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Early termination.
Units Other Than Participants: Restoration type
Groups:
- Restoration With Surefil One Hybrid Composite: In a split-mouth design, subjects were randomly assigned to restoration with Surefil one hybrid composite in either the left or the right upper quadrant.
  Restoration will be performed with Surefil one hybrid composite applied according to manufacturer's instruction and cured for 20 seconds with a LED lamp (Smartlamp Pro).
  Surefil one: Restorative material (Dentsply Sirona). Used for direct restoration of class V NCCL.
- Restoration With Venus Pearl Composite: In a split-mouth design, subjects were randomly assigned to restoration with Venus Pearl composite in either the left or the right upper quadrant.
  After the application of the adhesive system (iBond universal), the Venus Pearl composite will be layered on the cavity and cured for 20 seconds with a LED lamp Smartlamp Pro).
  Venus Pearl: Restorative material. Traditional paste composite employed in combination with iBond universal adhesive.
Period: Overall Study
Arm/Group | Restoration With Surefil One Hybrid Composite | Restoration With Venus Pearl Composite
Started | 16; 16 Restoration type | 16; 16 Restoration type
Completed | 16; 16 Restoration type | 16; 16 Restoration type
Not Completed | 0; 0 Restoration type | 0; 0 Restoration type

BASELINE CHARACTERISTICS:
Units Other Than Participants: Restoration type
Groups:
- Total: Total of all reporting groups
Arm/Group | Restoration With Surefil One Hybrid Composite | Restoration With Venus Pearl Composite | Total
Number analyzed (Participants) | 16 | 16 | 16
Number analyzed (Restoration type) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 10 | 10 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Restorative Quality
Description: The restorations will be evaluated using the World Dental Federation (FDI) criteria.
Time Frame: At 36 months follow-up.
Population: Premature termination of study.
Groups:
- Restoration With Surefil One Hybrid Composite: Restoration will be performed with Surefil one hybrid composite applied according to manufacturer's instruction and cured for 20 seconds with a LED lamp (Smartlamp Pro).
  Surefil one: Restorative material (Dentsply Sirona). Used for direct restoration of class V NCCL.
- Restoration With Venus Pearl Composite: After the application of the adhesive system (iBond universal), the Venus Pearl composite will be layered on the cavity and cured for 20 seconds with a LED lamp Smartlamp Pro).
  Venus Pearl: Restorative material. Traditional paste composite employed in combination with iBond universal adhesive.
Arm/Group | Restoration With Surefil One Hybrid Composite | Restoration With Venus Pearl Composite
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Assessment of Restorative Quality
Description: The restorations will be evaluated using the United States Public Health Service (USPHS) criteria.
Time Frame: At 36 months follow-up
Population: Premature termination of study.
Arm/Group | Restoration With Surefil One Hybrid Composite | Restoration With Venus Pearl Composite
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Assessment of Restorative Quality
Description: The restorations will be evaluated using the FDI criteria.
Time Frame: At 6, 12 and 24 months follow-up
Reporting Status: Not Posted

4. Secondary Outcome: Assessment of Restorative Quality
Description: The restorations will be evaluated using the USPHS criteria.
Time Frame: At 6, 12 and 24 months follow-up
Reporting Status: Not Posted

5. Secondary Outcome: Assessment of Aesthetics
Description: The aesthetic integration of the restoration will be evaluated by two experienced and blinded operators following the aesthetic criteria of the FDI.
Time Frame: At 6, 12, 24 and 36 months follow-up
Reporting Status: Not Posted

6. Secondary Outcome: Level of Pain
Description: Sensitivity index: thermal yes/no, if yes then Visual Analogue Scale (VAS) index for level of pain. Air yes/no, if yes then VAS index for level of pain.
Time Frame: At 6, 12, 24 and 36 months follow-up
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Time Needed to Perform the Restoration
Description: The time needed to perform the restorations will be compared between the groups.
Time Frame: Day 0
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 16 months.
Arm/Group | Restoration With Surefil One Hybrid Composite | Restoration With Venus Pearl Composite
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT05751382/Prot_SAP_000.pdf